CLINICAL TRIAL: NCT01559883
Title: Study on Thrombosis Therapy in German Cancer Patients
Status: Completed | Type: Observational
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: DE-Thrombose-NIS-2012
Record Dates: First submitted 2012-03-01; First posted 2012-03-21 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2013-11

CONDITIONS: Cancer; Deep Vein Thrombosis; Pulmonary Embolism
Keywords: cancer; thrombosis; pulmonary embolism; anticoagulation; low molecular weight heparin
MeSH Terms: conditions — Neoplasms; Venous Thrombosis; Pulmonary Embolism; Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- all eligible patients: there is only 1 Cohort in which all patients participating in this NIS are included
  Interventions: Other: no intervention is being made

INTERVENTIONS:
Other: no intervention is being made — This is a Non-Interventional Study (NIS)

SUMMARY:
The study aims to document the flow of German patients with cancer and acute deep vein thrombosis from first visit to diagnosis and treatment, the applied diagnostic procedures, and therapy modalities.

ELIGIBILITY:
Inclusion Criteria:

* patient with cancer and acute deep vein thrombosis and/or pulmonary embolism

Exclusion Criteria:

* life expectancy less that 6 months
* age less that 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer patient with acute deep vein throbosis/ pulmonary embolism in ambulatory oncology care/practice
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2012-02; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
treatment time on low molecular weight heparin | 1 year

SECONDARY OUTCOMES:
patient pathways | 1 year
  data collection on patient pathway: who is the referring physician, physician who diagnoses deep vein thrombosis (DVT)
risk factors for DVT | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Axel Matzdorff, Prof.Dr., Principal Investigator — Caritasklinikum Saarbrücken, St. Theresia
Locations (1):
- Prof. Dr. Axel Matzdorff, Saarbrücken, Saarland, Germany